CLINICAL TRIAL: NCT02841189
Title: King Vision Video Laryngoscope aBlade System for Use in Children
Brief Title: King Vision Video Laryngoscope Ambu (aBlade) System for Use in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Collaborators: King Systems Corporation (Industry)
Responsible Party: Principal Investigator, Nicole Horn, pediatric anesthesiologist, Indiana University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 1409265337
Record Dates: First submitted 2016-05-13; First posted 2016-07-22 (Estimated); Results first posted 2020-06-02 (Actual); Last update posted 2020-06-02 (Actual); Status verified 2020-05

CONDITIONS: Pediatric Anesthesia; King Vision Video Laryngoscope Intubation

ARMS (1):
- Video laryngoscope intubation (Other): The King Vision Video Laryngoscope will be used for intubation
  Interventions: Device: King Vision video Laryngoscope

INTERVENTIONS:
Device: King Vision video Laryngoscope — The King Vision video laryngoscope (Ambu) will be used for tracheal intubation.
  Other Names: Ambu

SUMMARY:
This is a single center trial to evaluate the performance of the King Vision video laryngoscope in pediatric patients between the ages of one month and 10 years of age. If the performance is satisfactory, this device may become a standard laryngoscope for tracheal intubation in elective and emergent tracheal intubations.

ELIGIBILITY:
Inclusion Criteria:

1. All children between the ages of 1 month to 10 years with a normal preoperative airway examination
2. Scheduled for a surgical procedure that requires tracheal intubation shall be included.

Exclusion Criteria:

1. Patients that will be excluded are those with an airway examination or previous anesthesia history that suggests difficulty with mask ventilation.

Ages: 1 Month to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2014-12; Primary Completion 2017-11-07 (Actual); Study Completion 2017-11-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicole Horn, MD, Principal Investigator — Riley Hospital
Locations (1):
- Riley Hospital for Children at IU Health, Indianapolis, Indiana, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Ease of Endotracheal Tube Passage: Intubations rated as "easy" and answers collected yes or no. s
Period: Overall Study
Arm/Group | Ease of Endotracheal Tube Passage
Started | 100
Completed | 65
Not Completed | 35

BASELINE CHARACTERISTICS:
Groups:
- Participants: Participant details
Arm/Group | Participants
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 100
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 45
  Male | 55
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Ease of Endotracheal Intubation
Description: Ease of endotracheal intubation
Time Frame: During intubation
Measure: Number; unit: participants
Groups:
- Ease of Endotracheal Tube Passage: Intubations rated as "easy" with data score of 1 or 2
Arm/Group | Ease of Endotracheal Tube Passage
Number analyzed (Participants) | 65
participants | 65

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- Adverse Event Participants: Adverse event affecting participant details
Arm/Group | Adverse Event Participants
All-Cause Mortality (participants affected / at risk) | 0/65
Serious Adverse Events (participants affected / at risk) | 0/65
Other Adverse Events (participants affected / at risk) | 0/65

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Study Protocol (2016-03-28): https://cdn.clinicaltrials.gov/large-docs/89/NCT02841189/Prot_SAP_000.pdf
  • Informed Consent Form (2016-05-18): https://cdn.clinicaltrials.gov/large-docs/89/NCT02841189/ICF_001.pdf
  • Statistical Analysis Plan: Data collection Sheet (2015-09-14): https://cdn.clinicaltrials.gov/large-docs/89/NCT02841189/SAP_002.pdf